CLINICAL TRIAL: NCT05547867
Title: Elbow Heterotopic Ossifications Associated With Radial Head Prosthesis: Risk and Prognostic Factors
Brief Title: Elbow Heterotopic Ossifications Associated With Radial Head Prosthesis
Acronym: Prosthesis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-RAD-2022-52
Record Dates: First submitted 2022-09-11; First posted 2022-09-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2023-09

CONDITIONS: Radial Head Fracture
MeSH Terms: conditions — Radial Head and Neck Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Radial head prosthesis — Radial head arthroplasty in comminuted radial head fractures.

SUMMARY:
Elbow heterotopic ossification (EHO) is described as the formation of ectopic bone in tissues not supposed to around elbow. The EHO physiopathology, yet not clarified, has been suggested to be a multifactorial process in which immune system, inflammatory response, CNS and tissue expressed proteins after severe trauma boost hyperactive metabolically bone with no periosteal layer. Consistent with that, EHO has been widely related to elbow trauma, including bone, ligament, muscle or joint; iatrogenic trauma, including epicondylectomy or elbow arthroplasty; neural injuries or burns. Clinical manifestations of EHO has been reported as limited range of motion (ROM), muscle, nerve or joint pain, stiffness and ankylosis all of them leading to upper extremity disfucntion. Prevalence of EHO can range from 3%-45% depending on degree of elbow injury. To our knowledge, prevalence of EHO among radial head fractures had not been assessed previously.

DETAILED DESCRIPTION:
Prevention of EHO has been proposed to be managed with a range of nonsurgical treatment options such as: radiotherapy, NSAIDS and biphosphonate. However, none of them had become clear effective above others, and only surgical excision of EHO had become a reliable option to overcome its associated limitations in elbow motion. Classic approaches suggested delayed surgery until maturity of heterotopic bone, however recent literature suggest early excisions of immature ossification to obtain favorable functional results.

Several studies have investigated risk factors of EHO regarding the high patient burden and health costs to which is associated, however, few published data exists about prevalence and risk factors of EHO after radial head arthroplasty.

Our aim is to assess the prevalence and predictor factors that can lead to EHO after radial arthroplasty in order to be able to predict and apply early preventive treatment to improve postoperative functional outcomes among patients with severe radial head fractures.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 18-85 years-old
* Comminuted radial head fractures treated with radial head arthroplasty

Exclusion Criteria:

* Younger than 18 years; Older than 85 years
* History of previous elbow injuries or operations.
* Pathologic fractures
* Infections

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The present study will include consecutive patients admitted to our hospital Hospital de la Santa Creu i Sant Pau (Barcelona, Spain) elected for radial head arthroplasty due to elbow fractures from 2010 to 2020. All patients will be included retrospectively through our hospital patient electronic health records.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-09-12 (Actual); Primary Completion 2024-06-10 (Estimated); Study Completion 2024-09-09 (Estimated)

PRIMARY OUTCOMES:
Prevalence of EHO | 12 months
  Assess prevalence of EHO after radial head arthroplasty in anteroposterior and lateral radiographs.
Average size of EHO | 12 months
  Size of EHO (measure in mm) in X-rays.
Site of EHO in elbow | 12 months
  Location of EHO in elbow anteroposterior and lateral X-rays (anterior, posterior, medial, lateral).
Osteopenia of the capitellum | 12 months
  The radiographs of the elbow will be review for osteopenia of the capitellum, and graded as none, mild, moderate, or severe according to the system of Lamas et al. (2011).
Degenerative changes of the elbow | 12 months
  In anteroposterior and lateral X-rays. For the degree of degenerative change of the elbow, classified as Grade 0 (normal joint), Grade 1 (slight joint, space narrowing and minimum osteophyte formation), Grade 2 (moderate joint space narrowing and moderate osteophyte formation), or Grade 3 (severe degenerative changes with gross destruction of the joint) according to the system of Broberg and Morrey (1986).

SECONDARY OUTCOMES:
Radial head fracture and associated elbow lesions | 12 months
  We classified the radial head fracture by Mason´s classification with the Johnston modification (Fracture types I, II, III, IV) (1954).

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Lamas, MD Ph D, Principal Investigator — HSCSP
Locations (2):
- Spain (2):
  - Claudia Erika Delgado Espinoza, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona

IPD SHARING:
Plan to Share IPD: No
Protocol for the collection of radiological data and possible risk and prognostic factors associated with the presence of EHO in radial head arthroplasty.

REFERENCES:
- [Result] Barfield WR, Holmes RE, Hartsock LA. Heterotopic Ossification in Trauma. Orthop Clin North Am. 2017 Jan;48(1):35-46. doi: 10.1016/j.ocl.2016.08.009. Epub 2016 Oct 28. PMID 27886681
- [Result] Qazi S, Reynolds J, Abdelfattah H, Thoder J. Heterotopic Ossification of the Elbow: A Literature Review. J Adv Med Med Res. August 2019:1-10. doi:10.9734/JAMMR/2019/V30I630207
- [Result] Summerfield SL, DiGiovanni C, Weiss AP. Heterotopic ossification of the elbow. J Shoulder Elbow Surg. 1997 May-Jun;6(3):321-32. doi: 10.1016/s1058-2746(97)90025-2. No abstract available. PMID 9219141
- [Result] Agarwal S, Loder S, Levi B. Heterotopic Ossification Following Upper Extremity Injury. Hand Clin. 2017 May;33(2):363-373. doi: 10.1016/j.hcl.2016.12.013. PMID 28363301
- [Result] Robinson PM, MacInnes SJ, Stanley D, Ali AA. Heterotopic ossification following total elbow arthroplasty: a comparison of the incidence following elective and trauma surgery. Bone Joint J. 2018 Jun 1;100-B(6):767-771. doi: 10.1302/0301-620X.100B6.BJJ-2017-0535.R2. PMID 29855240
- [Result] Baldwin K, Hosalkar HS, Donegan DJ, Rendon N, Ramsey M, Keenan MA. Surgical resection of heterotopic bone about the elbow: an institutional experience with traumatic and neurologic etiologies. J Hand Surg Am. 2011 May;36(5):798-803. doi: 10.1016/j.jhsa.2011.01.015. Epub 2011 Apr 2. PMID 21458925
- [Result] KAPICIOĞLU M, SAĞLAM Y, ERŞEN A, ATALAR AC, DEMİRHAN M, DURMAZ H. Does Resection of Heterotopic Ossification of the Elbow Result in Satisfactory Functional Outcomes? Bezmialem Sci. 2019;7(2):124-131. doi:10.14235/bas.galenos.2018.2467
- [Result] Foruria AM, Augustin S, Morrey BF, Sanchez-Sotelo J. Heterotopic ossification after surgery for fractures and fracture-dislocations involving the proximal aspect of the radius or ulna. J Bone Joint Surg Am. 2013 May 15;95(10):e66. doi: 10.2106/JBJS.K.01533. PMID 23677367
- [Result] van Kampen PJ, Martina JD, Vos PE, Hoedemaekers CW, Hendricks HT. Potential risk factors for developing heterotopic ossification in patients with severe traumatic brain injury. J Head Trauma Rehabil. 2011 Sep-Oct;26(5):384-91. doi: 10.1097/HTR.0b013e3181f78a59. PMID 21321512
- [Result] Salazar D, Golz A, Israel H, Marra G. Heterotopic ossification of the elbow treated with surgical resection: risk factors, bony ankylosis, and complications. Clin Orthop Relat Res. 2014 Jul;472(7):2269-75. doi: 10.1007/s11999-014-3591-0. Epub 2014 Apr 8. PMID 24711127
- [Result] Ploumis A, Belbasis L, Ntzani E, Tsekeris P, Xenakis T. Radiotherapy for prevention of heterotopic ossification of the elbow: a systematic review of the literature. J Shoulder Elbow Surg. 2013 Nov;22(11):1580-8. doi: 10.1016/j.jse.2013.07.045. PMID 24138821
- [Result] Garland DE. A clinical perspective on common forms of acquired heterotopic ossification. Clin Orthop Relat Res. 1991 Feb;(263):13-29. PMID 1899635
- [Result] Suito M, Yuzuriha S, Iwasawa M, Yanagisawa D, Kinjo Y, Takashimizu I, Hoshino Y. Therapeutic strategies for elbow ankylosis due to heterotopic ossification in patients with severe burns. JPRAS Open. 2018 Jul 5;17:24-30. doi: 10.1016/j.jpra.2018.06.004. eCollection 2018 Sep. PMID 32158828
- [Result] Wiggers JK, Helmerhorst GT, Brouwer KM, Niekel MC, Nunez F, Ring D. Injury complexity factors predict heterotopic ossification restricting motion after elbow trauma. Clin Orthop Relat Res. 2014 Jul;472(7):2162-7. doi: 10.1007/s11999-013-3304-0. PMID 24078170
- [Result] Abrams GD, Bellino MJ, Cheung EV. Risk factors for development of heterotopic ossification of the elbow after fracture fixation. J Shoulder Elbow Surg. 2012 Nov;21(11):1550-4. doi: 10.1016/j.jse.2012.05.040. Epub 2012 Sep 2. PMID 22947234
- [Result] Bauer AS, Lawson BK, Bliss RL, Dyer GS. Risk factors for posttraumatic heterotopic ossification of the elbow: case-control study. J Hand Surg Am. 2012 Jul;37(7):1422-9.e1-6. doi: 10.1016/j.jhsa.2012.03.013. Epub 2012 May 1. PMID 22551954
- [Result] Hong CC, Nashi N, Hey HW, Chee YH, Murphy D. Clinically relevant heterotopic ossification after elbow fracture surgery: a risk factors study. Orthop Traumatol Surg Res. 2015 Apr;101(2):209-13. doi: 10.1016/j.otsr.2014.10.021. Epub 2015 Feb 18. PMID 25701160
- [Result] Schnetzke M, Porschke F, Hoppe K, Studier-Fischer S, Gruetzner PA, Guehring T. Outcome of Early and Late Diagnosed Essex-Lopresti Injury. J Bone Joint Surg Am. 2017 Jun 21;99(12):1043-1050. doi: 10.2106/JBJS.16.01203. PMID 28632594
- [Result] Broberg MA, Morrey BF. Results of delayed excision of the radial head after fracture. J Bone Joint Surg Am. 1986 Jun;68(5):669-74. PMID 3722222
- [Result] Lamas C, Castellanos J, Proubasta I, Dominguez E. Comminuted radial head fractures treated with pyrocarbon prosthetic replacement. Hand (N Y). 2011 Mar;6(1):27-33. doi: 10.1007/s11552-010-9282-8. Epub 2010 Jun 15. PMID 22379435